CLINICAL TRIAL: NCT01124669
Title: BRAF, KRAS and EGFR Mutation Detection in Non-Small Cell Lung Cancer Patients Treated With Sorafenib Monotherapy
Brief Title: Biomarkers in Blood Samples From Patients With Refractory Non-Small Cell Lung Cancer Previously Treated With Sorafenib Tosylate
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000670998; ECOG-E2501T2
Record Dates: First submitted 2010-05-14; First posted 2010-05-17 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: DNA analysis
Genetic: mutation analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in blood samples from patients with refractory non-small cell lung cancer previously treated with sorafenib tosylate.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the mutation rates of BRAF, KRAS, and EGFR in patients with non-small cell lung cancer treated with sorafenib tosylate on protocol ECOG-2501.
* To determine the association between BRAF, KRAS, or EGFR mutation status and clinical benefits in patients treated with this regimen.

OUTLINE: This is a multicenter study.

DNA is isolated from archived plasma samples and analyzed for BRAF, KRAS, and EGFR mutations.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of refractory non-small cell lung cancer
* Received sorafenib tosylate on protocol ECOG-E2501
* Available blood specimens

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patients enrolled on E2501
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-06-13 (Actual); Primary Completion 2010-07-13 (Actual); Study Completion 2010-07-13 (Actual)

PRIMARY OUTCOMES:
Mutation rate of sorafenib tosylate-target gene BRAF, and its upstream proteins KRAS and EGFR | 1 mont
Association between BRAF, KRAS, and EGFR mutation status and clinical benefits (stable disease or partial response) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chung, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center